CLINICAL TRIAL: NCT01847547
Title: Comparative Effectiveness of Oral Anticoagulants: A Cohort Study
Brief Title: Comparative Effectiveness of Oral Anticoagulants
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.157
Record Dates: First submitted 2013-04-18; First posted 2013-05-07 (Estimated); Results first posted 2014-05-19 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Dabigatran
- Warfarin

SUMMARY:
This cohort study plans to identify initiators of oral anticoagulants using electronic claims data from a commercial insurance database to quantify associations between anticoagulant choice (warfarin and dabigatran) and the occurrence of selected outcomes in patients with non-valvular atrial fibrillation at risk for stroke.

ELIGIBILITY:
Inclusion criteria:

* A recorded diagnosis of atrial fibrillation (AF).
* Initiation of anticoagulant medication (dabigatran or warfarin).
* At least 18 years of age on the date of anticoagulant initiation CHA2DS2-VASc-Score >=1

Exclusion criteria:

* Patients with missing or ambiguous age or sex information
* Patients with documented evidence of valvular disease
* Patients with less than 12 months enrolment in the UnitedHealth Research Database preceding the date of anticoagulant initiation
* Patients with prior use of any oral anticoagulant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age and older with non-valvular AF initiating oral anticoagulation therapy
Sampling Method: Non-Probability Sample
Enrollment: 5982 (Actual)
Dates: Start 2013-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an observational study. Patients were not actively recruited in this study. The data source was the UnitedHealth database.
Pre-assignment Details: 11882 patients fulfilled the in- and ex-clusion criteria. Only 5982 patients remained after matching on the Propensity Score.
Groups:
- Dabigatran: Propensity score matched patients starting treatment with dabigatran
- Warfarin: Propensity score matched patients starting treatment with warfarin
Period: Overall Study
Arm/Group | Dabigatran | Warfarin
Started | 2991 | 2991
Completed | 2991 | 2991
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This initial cohort study includes matched treatment groups of 2,991 patients with non-valvular atrial fibrillation who initiated dabigatran and 2,991 patients who initiated warfarin that were drawn from a pool of 11,882 eligible initiators. These first feasibility data are limited by a small sample size.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran | Warfarin | Total
Number analyzed (Participants) | 2991 | 2991 | 5982
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.86 (10.99) | 63.26 (11.04) | 63.60 (11.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 943 | 877 | 1820
  Male | 2048 | 2114 | 4162

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Stroke
Description: Events during follow-up (October 2010- 30 June 2012) were identified using ICD 9 codes.
Time Frame: From treatment initiation until end of follow-up; up to 20 months
Population: Hazard ratios and confidence intervals were estimated for patients starting dabigatran or warfarin after matching on the propensity score.
Measure: Number; unit: events per 1000 person years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 2991 | 2991
events per 1000 person years | 29.09 | 31.59
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; These current feasibility data are limited by a small sample size, short follow up, and few outcome events resulting in wide 95% confidence intervals. At this early stage, no comparative conclusions are possible. Future data with an increased number of patients are planned; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 1.05, 95% CI [0.64 to 1.70] — Cox Proportional Hazard's regression following propensity score matching

2. Primary Outcome: Incidence Rate of Major Bleeding
Description: Events during follow-up (October 2010- 30 June 2012) were identified using ICD 9 and procedure codes.
Time Frame: From treatment initiation until end of follow-up; up to 20 months
Population: as for outcome 1
Measure: Number; unit: events per 1000 person years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 2991 | 2991
events per 1000 person years | 60.00 | 66.72
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 0.97, 95% CI [0.69 to 1.36] — Cox Proportional Hazard's regression following propensity score matching

3. Secondary Outcome: Incidence Rate of Myocardial Infarction
Description: Events during follow-up (October 2010- 30 June 2012) were identified using ICD 9 codes.
Time Frame: From treatment initiation until end of follow-up; up to 20 months
Population: as for outcome 1
Measure: Number; unit: events per 1000 person years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 2991 | 2991
events per 1000 person years | 16.90 | 14.73
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 1.24, 95% CI [0.62 to 2.45] — Cox Proportional Hazard's regression following propensity score matching

4. Secondary Outcome: Incidence Rate of Venous Thromboembolism
Description: Events during follow-up (October 2010- 30 June 2012) were identified using ICD 9 codes.
Time Frame: From treatment initiation until end of follow-up; up to 20 months
Population: as for outcome 1
Measure: Number; unit: events per 1000 person years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 2991 | 2991
events per 1000 person years | 8.83 | 34.79
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 0.29, 95% CI [0.15 to 0.59] — Cox Proportional Hazard's regression following propensity score matching

5. Secondary Outcome: Incidence Rate of Deep Vein Thrombosis
Description: Events during follow-up (October 2010- 30 June 2012) were identified using ICD 9 codes.
Time Frame: From treatment initiation until end of follow-up; up to 20 months
Population: as for outcome 1
Measure: Number; unit: events per 1000 person years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 2991 | 2991
events per 1000 person years | 7.23 | 27.35
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; These current feasibility data are limited by a small sample size, short follow up, and few outcome events resulting in wide 95% confidence intervals. At this early stage, no comparative conclusions are possible; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 0.31, 95% CI [0.15 to 0.67] — Cox Proportional Hazard's regression following propensity score matching

6. Secondary Outcome: Incidence Rate of Pulmonary Embolism
Description: Events during follow-up (October 2010- 30 June 2012) were identified using ICD 9 codes.
Time Frame: From treatment initiation until end of follow-up; up to 20 months
Population: as for outcome 1
Measure: Number; unit: events per 1000 person years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 2991 | 2991
events per 1000 person years | 3.21 | 13.65
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 0.27, 95% CI [0.09 to 0.84] — Cox Proportional Hazard's regression following propensity score matching

7. Secondary Outcome: Incidence Rate of Major Lower Gastrointestinal Bleeding
Description: Events during follow-up (October 2010- 30 June 2012) were identified using ICD 9 codes.
Time Frame: From treatment initiation until end of follow-up; up to 20 months
Population: as for outcome 1
Measure: Number; unit: events per 1000 person years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 2991 | 2991
events per 1000 person years | 35.52 | 30.57
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 1.25, 95% CI [0.78 to 2.01] — Cox Proportional Hazard's regression following propensity score matching

8. Secondary Outcome: Incidence Rate of Major Urogenital Bleeding
Description: Events during follow-up (October 2010- 30 June 2012) were identified using ICD 9 codes.
Time Frame: From treatment initiation until end of follow-up; up to 20 months
Population: as for outcome 1
Measure: Number; unit: events per 1000 person years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 2991 | 2991
events per 1000 person years | 0.0 | 0.0

9. Secondary Outcome: Incidence Rate of Major Other Bleeding
Description: Events during follow-up (October 2010- 30 June 2012) were identified using ICD 9 codes.
Time Frame: From treatment initiation until end of follow-up; up to 20 months
Population: as for outcome 1
Measure: Number; unit: events per 1000 person years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 2991 | 2991
events per 1000 person years | 32.25 | 46.41
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 0.74, 95% CI [0.48 to 1.14] — Cox Proportional Hazard's regression following propensity score matching

10. Secondary Outcome: Incidence Rate of Transient Ischemic Attack
Description: Events during follow-up (October 2010- 30 June 2012) were identified using ICD 9 codes.
Time Frame: From treatment initiation until end of follow-up; up to 20 months
Population: as for outcome 1
Measure: Number; unit: events per 1000 person years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 2991 | 2991
events per 1000 person years | 11.27 | 12.61
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 1.01, 95% CI [0.47 to 2.20] — Cox Proportional Hazard's regression following propensity score matching

11. Secondary Outcome: Incidence Rate of Major Upper Gastrointestinal Bleeding
Description: Events during follow-up (October 2010- 30 June 2012) were identified using ICD 9 and procedure codes.
Time Frame: From treatment initiation until end of follow-up; up to 20 months
Population: as for outcome 1
Measure: Number; unit: events per 1000 person years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 2991 | 2991
events per 1000 person years | 4.82 | 7.34
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; These current feasibility data are limited by a small sample size, short follow up, and very few outcome events resulting in wide 95% confidence intervals. At this early stage, no comparative conclusions are possible. Future data with an increased number of patients are planned; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 0.65, 95% CI [0.21 to 1.98] — Cox Proportional Hazard's regression following propensity score matching

12. Secondary Outcome: Incidence Rate of Stroke or Systemic Embolism
Description: Events during follow-up (October 2010- 30 June 2012) were identified using ICD 9 codes.
Time Frame: From treatment initiation until end of follow-up; up to 20 months
Population: as for outcome 1
Measure: Number; unit: events per 1000 person years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 2991 | 2991
events per 1000 person years | 39.73 | 60.38
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 0.74, 95% CI [0.50 to 1.08] — Cox Proportional Hazard's regression following propensity score matching

13. Secondary Outcome: Incidence Rate of Systemic Embolism
Description: Events during follow-up (October 2010- 30 June 2012) were identified using ICD 9 codes.
Time Frame: From treatment initiation until end of follow-up; up to 20 months
Population: as for outcome 1
Measure: Number; unit: events per 1000 person years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 2991 | 2991
events per 1000 person years | 11.27 | 30.55
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 0.40, 95% CI [0.21 to 0.76] — Cox Proportional Hazard's regression following propensity score matching

14. Secondary Outcome: Incidence Rate of Ischemic Stroke
Description: Events during follow-up (October 2010- 30 June 2012) were identified using ICD 9 codes.
Time Frame: From treatment initiation until end of follow-up; up to 20 months
Population: as for outcome 1
Measure: Number; unit: events per 1000 person years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 2991 | 2991
events per 1000 person years | 27.40 | 32.71
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 0.95, 95% CI [0.58 to 1.55] — Cox Proportional Hazard's regression following propensity score matching

15. Secondary Outcome: Incidence Rate of Hemorrhagic Stroke
Description: Events during follow-up (October 2010- 30 June 2012) were identified using ICD 9 codes.
Time Frame: From treatment initiation until end of follow-up; up to 20 months
Population: as for outcome 1
Measure: Number; unit: events per 1000 person years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 2991 | 2991
events per 1000 person years | 4.02 | 3.14
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 1.36, 95% CI [0.32 to 5.72] — Cox Proportional Hazard's regression following propensity score matching

16. Secondary Outcome: Incidence Rate of Stroke Uncertain Classification
Description: Events during follow-up (October 2010- 30 June 2012) were identified using ICD 9.
Time Frame: From treatment initiation until end of follow-up; up to 20 months
Population: as for outcome 1
Measure: Number; unit: events per 1000 person years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 2991 | 2991
events per 1000 person years | 20.98 | 14.70
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 1.60, 95% CI [0.83 to 3.08] — Cox Proportional Hazard's regression following propensity score matching

17. Secondary Outcome: Incidence Rate of Major Intracranial Bleeding
Description: Events during follow-up (October 2010- 30 June 2012) were identified using ICD 9 codes.
Time Frame: From treatment initiation until end of follow-up; up to 20 months
Population: as for outcome 1
Measure: Number; unit: events per 1000 person years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 2991 | 2991
events per 1000 person years | 9.65 | 7.34
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 1.45, 95% CI [0.57 to 3.70] — Cox Proportional Hazard's regression following propensity score matching

18. Secondary Outcome: Incidence Rate of Major Extracranial Bleeding
Description: Events during follow-up (October 2010- 30 June 2012) were identified using ICD 9 and procedure codes.
Time Frame: From treatment initiation until end of follow-up; up to 20 months
Population: as for outcome 1
Measure: Number; unit: events per 1000 person years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 2991 | 2991
events per 1000 person years | 56.70 | 63.53
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 0.95, 95% CI [0.67 to 1.35] — Cox Proportional Hazard's regression following propensity score matching

19. Secondary Outcome: Incidence Rate of Major Gastrointestinal Bleeding
Description: Events during follow-up (October 2010- 30 June 2012) were identified using ICD 9 and procedure codes.
Time Frame: From treatment initiation until end of follow-up; up to 20 months
Population: as for outcome 1
Measure: Number; unit: events per 1000 person years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 2991 | 2991
events per 1000 person years | 37.14 | 31.63
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 1.26, 95% CI [0.79 to 2.01] — Cox Proportional Hazard's regression following propensity score matching

ADVERSE EVENTS:
Time Frame: Up to 20 months
Arm/Group | Dabigatran | Warfarin
Serious Adverse Events (participants affected / at risk) | 0/2991 | 0/2991
Other Adverse Events (participants affected / at risk) | 0/2991 | 0/2991

LIMITATIONS AND CAVEATS:
These first data are limited by small sample size, short follow up, few events resulting in wide confidence intervals. No comparative conclusions are possible. After the feasibility analysis future analysis will increase patient numbers and follow up

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No